CLINICAL TRIAL: NCT05585320
Title: A Phase 1/2a, Open-Label, Multicenter, Nonrandomized, Safety and Anti-tumor Activity Study of IMM-1-104, a Novel Oral Dual MEK1/2 Inhibitor in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Phase 1/2a Study of IMM-1-104 in Participants With Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immuneering Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM1104-101
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; Pancreatic Adenocarcinoma; Malignant Melanoma (Cutaneous); Non-small Cell Lung Cancer (NSCLC)
Keywords: pan-RAS; KRAS; NRAS; HRAS; Targeted therapy; Metastatic cancer; Advanced cancer; RAS; Adenocarcinoma; MEK; Dual MEK; MEK 1/2; Mitogen-Activated Protein Kinase (MAPK); G12A; G12C; G12D; G12F; G12R; G12S; G12V; G13C; G13D; G13R; Q61H; Q61K; Q61L; Q61R; A146T; A146V; K117N
MeSH Terms: conditions — Melanoma, Cutaneous Malignant; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Adenocarcinoma | interventions — dabrafenib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- IMM-1-104 monotherapy (Treatment Group A) (Experimental): IMM-1-104 monotherapy for first/second line pancreatic adenocarcinoma; first/second/third line melanoma; or second/third line non small cell lung cancer
  Interventions: Drug: IMM-1-104 Monotherapy (Treatment Group A)
- IMM-1-104 in combination with mGnP (Treatment Group B) (Experimental): IMM-1-104 in combination with modified gemcitabine and nab-paclitaxel (mGnP) for first line pancreatic adenocarcinoma
  Interventions: Drug: IMM-1-104 + modified Gemcitabine/nab-Paclitaxel (Treatment Group B)
- IMM-1-104 in combination with mFFX (Treatment Group C) (Experimental): IMM-1-104 in combination with modified FOLFIRINOX (mFFX) for first line pancreatic adenocarcinoma
  Interventions: Drug: IMM-1-104 + modified FOLFIRINOX (Treatment Group C)
- IMM-1-104 in combination with dabrafenib (Treatment Group D) (Experimental): IMM-1-104 in combination with dabrafenib for second/third line post-IO melanoma with BRAF mutation
  Interventions: Drug: IMM-1-104 + dabrafenib (Treatment Group D)
- IMM-1-104 in combination with pembrolizumab (Treatment Group E) (Experimental): IMM-1-104 in combination with pembrolizumab for second/third line post-IO melanoma
  Interventions: Drug: IMM-1-104 + pembrolizumab (Treatment Group E)

INTERVENTIONS:
Drug: IMM-1-104 Monotherapy (Treatment Group A) — Once-daily, oral IMM-1-104 dose administered in 28-day cycles until treatment discontinuation criteria are met
  Other Names: IMM-1-104
  Arms: IMM-1-104 monotherapy (Treatment Group A)
Drug: IMM-1-104 + modified Gemcitabine/nab-Paclitaxel (Treatment Group B) — Once-daily, oral IMM-1-104 dose administered in 28-day cycles in combination with intravenous infusions of gemcitabine and nab-paclitaxel until treatment discontinuation criteria are met.
  Gemcitabine will be administered at a dose of 1000 mg/m^2 nab-Paclitaxel will be administered at a dose of 125 mg/m^2
  Other Names: IMM-1-104 + mGnP
  Arms: IMM-1-104 in combination with mGnP (Treatment Group B)
Drug: IMM-1-104 + modified FOLFIRINOX (Treatment Group C) — Once-daily, oral IMM-1-104 dose administered in 28-day cycles in combination with intravenous infusions of modified FOLFIRNOX until treatment discontinuation criteria are met.
  FOLFIRINOX will be administered as follows:
  Folinic Acid will be administered at 400 mg/m^2 Fluorouracil will be administered at 2400 mg/m^2 Irinotecan will be administered at 150 mg/m^2 Oxaliplatin will be administered at 85 mg/m^2
  Other Names: IMM-1-104 + mFFX
  Arms: IMM-1-104 in combination with mFFX (Treatment Group C)
Drug: IMM-1-104 + dabrafenib (Treatment Group D) — Once-daily, oral IMM-1-104 dose administered in 28-day cycles in combination with twice daily oral dose of dabrafenib until treatment discontinuation criteria are met. Dabrafenib will be administered at a dose of 150mg daily (75mg twice daily).
  Other Names: IMM-1-104 + dabrafenib
  Arms: IMM-1-104 in combination with dabrafenib (Treatment Group D)
Drug: IMM-1-104 + pembrolizumab (Treatment Group E) — Once-daily, oral IMM-1-104 dose administered in 28-day cycles in combination with intravenous infusions of pembrolizumab in sequence or concurrently depending on the enrolled cohort (two sub cohorts) until treatment discontinuation criteria are met. Pembrolizumab will be administered at a dose of 400mg.
  Other Names: IMM-1-104 + pembro
  Arms: IMM-1-104 in combination with pembrolizumab (Treatment Group E)

SUMMARY:
This is an open-label, dose-exploration and expansion study to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of IMM-1-104 when administered as monotherapy or in combination with approved agents in participants with RAS-mutated or RAS/MAPK activated advanced or metastatic solid tumors. The dose exploration will identify the candidate recommended Phase 2 candidate optimal dose of IMM-1-104 to further explore the anti-tumor activity of IMM-1-104 as monotherapy and in combination with approved agents in multiple Phase 2a proof-of-concept cohorts in malignancies of interest.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥18 years of age
* Must have histologically or cytologically confirmed diagnosis as follows:

  1. Monotherapy Phase 1: A locally advanced unresectable or metastatic solid tumor malignancy that harbors a RAS (KRAS, NRAS, or HRAS) activating mutation.
  2. Monotherapy Phase 2a: A locally advanced unresectable or metastatic solid tumor malignancies: pancreatic ductal adenocarcinoma (PDAC), RAS-mutant melanoma, or RAS-mutant non-small cell lung cancer (NSCLC)
  3. Combination therapy (both phases): A locally advanced unresectable or metastatic PDAC
  4. Combination therapy Phase 2a, Treatment D: Second and third line participants with unresectable stage III or stage IV cutaneous melanoma with BRAF mutation. Must have progressed on or after treatment with an anti-PD-(L)1 monoclonal antibody as the most recent therapy. First day of study treatment must be more than 28 days but less than 12 weeks from the last dose of anti-PD-(L)1 mAb.
  5. Combination therapy Phase 2a, Treatment E: Second and third line participants with unresectable stage III or stage IV cutaneous melanoma. Must have progressed on or after treatment with an anti-PD-(L)1 monoclonal antibody as the most recent therapy. First day of study treatment must be more than 28 days but less than 12 weeks from the last dose of anti-PD-(L)1 mAb.
* Participants must be treatment naive or received prior systemic standard-of-care treatment as follows:

  1. Monotherapy Phase 1: received at least 1 line of systemic standard-of-care treatment for their advanced or metastatic disease
  2. Monotherapy Phase 2a:

     1. First-line PDAC participants will have received no previous systemic anti-cancer therapy. Second-line PDAC participants will have received no more than one prior systemic anti-cancer therapy.
     2. First-line melanoma participants will have received no previous systemic anti-cancer therapy. Second- and third-line participants will have received and failed one or two prior systemic anti-cancer therapies, respectively.
     3. NSCLC participants will have received at least one and no more than two previous lines of systemic therapy.
  3. Combination therapy (both phases): PDAC participants will have received no previous systemic anti-cancer therapy for their advanced or metastatic disease.
* Must have evidence of measurable disease (at least one target lesion) per RECIST v1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Inability to swallow oral medications
* Symptomatic, untreated, or actively progressing known central nervous system (CNS) metastases
* History or concurrent evidence of retinal vein occlusion (RVO) or current risk factors for RVO. History of serous retinopathy, retinal edema, or retinal pigment epithelial detachment (RPED)
* Impaired cardiovascular function or clinically significant cardiac disease
* History of rhabdomyolysis within 3 months prior to start of study treatment
* Active skin disorder requiring systemic treatment within 3 months prior to the start of study treatment
* Participants with active, uncontrolled autoimmune disease or participants actively being treated with tumor necrosis factor-alpha (TNF-alpha) inhibitors for management of their autoimmune disease are excluded
* Receipt of an allogeneic tissue/solid organ transplant
* Females who are pregnant, breastfeeding, or planning to become pregnant and males who plan to father a child while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Adverse Events | From treatment initiation through 30 days following the last IMM-1-104 dose
  Number of participants with adverse events
Phase 1: Dose-Limiting Toxicities | The first 21 days of study treatment
  Number of participants with dose-limiting toxicities
Phase 1: Recommended Phase 2 Candidate Optimal Dose | Initiation of study treatment through 21 days (up to approximately 18 months)
  Selection of candidate optimal dose to take forward into Ph2a
Phase 2a: Overall Response Rate | After up to 48 weeks (12 cycles) of study treatment
  The proportion of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR), based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Phase 1/2a: Maximum Observed Plasma Concentration of IMM-1-104 | After 12 weeks (3 Cycles) of study treatment
  Cmax
Phase 1/2a: Time to Reach Maximum Plasma Concentration of IMM-1-104 | After 12 weeks (3 Cycles) of study treatment
  Tmax
Phase 1/2a: Area Under Plasma Concentration (AUC) Time Curve of IMM-1-104 | After 12 weeks (3 Cycles) of study treatment
  AUC0-t
Phase 2a: Disease Control Rate (DCR) | After 16 weeks (4 Cycles) of study treatment
  The proportion of participants who have a best overall response (BOR) of stable disease (SD) or better
Phase 2a: Progression Free Survival (PFS) | Up to approximately 2 years
  The time interval between study treatment start and disease progression or death due to any cause.
Phase 2a: Duration of Response (DOR) | Up to approximately 2 years.
  The time interval between an assessment of partial response (PR) or better and disease progression or death due to any cause.
Phase 2a: Landmark 3-Month Survival | After 3 months of study participation.
  The proportion of participants who are still alive after three months on study.
Phase 2a: Landmark 6-Month Survival | After 6 months of study participation.
  The proportion of participants who are still alive after six months on study.
Phase 2a: Overall Survival (OS) | Up to approximately 2 Years
  The time interval between study treatment start and death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Vinny Hayreh, MD, Study Director — Immuneering Corporation
Locations (20):
- United States (20):
  - Mayo Clinic, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - University of California San Diego, San Diego, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mayo Clinic, Jacksonville, Florida
  - Florida Cancer Specialists and Research Institute, Lake Mary, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Weill Cornell Medicine, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Duke University Cancer Institute, Durham, North Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Oncology, Fairfax, Virginia
  - University of Wisconsin Clinical Science Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No